CLINICAL TRIAL: NCT06795633
Title: The Impact of a Holistic Care Program for High-Risk Pregnancies on Stress and Mental Health
Acronym: RGYBBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, Vice-dean, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RGYBBP
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: High-risk Pregnancy; Holistic Care; Stress; Prenatal Stress; Mental Health; Midwifery Support; Midwifery; Pregnancy; High-Risk Pregnancy School
Keywords: Holistic Care Practices; High-Risk Pregnancy; Midwifery; High-Risk Pregnancy School
MeSH Terms: conditions — Psychological Well-Being | interventions — Pregnancy, High-Risk

STUDY DESIGN:
Intervention Model Description: Intervention Group (50 participants): Received the holistic care program and routine midwifery care.
  Control Group (50 participants): Received routine midwifery care. Data were collected at two time points: a pre-test on the first day of group assignment and a post-test on the day of discharge.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group Applications: High-risk pregnant women admitted to the perinatology clinic and assigned to the intervention group participated in a Holistic Care Program for High-Risk Pregnancies in addition to the midwifery care provided at the clinic.
  Interventions: Other: Holistic Care Program for High-Risk Pregnancies
- Control Group (No Intervention): Control Group Applications: Routine midwifery care procedures followed in the perinatology clinic were applied to the control group.

INTERVENTIONS:
Other: Holistic Care Program for High-Risk Pregnancies — High-risk pregnant women admitted to the perinatology clinic participated in the Holistic Care Program for High-Risk Pregnancies in addition to the midwifery care provided in the clinic.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate the effects of the Holistic Care Program for High-Risk Pregnancies on the stress levels and mental health of pregnant women. Within this framework, the study seeks to examine the potential of the holistic care program to strengthen stress coping mechanisms, positively influence mental health, and enhance general health awareness among high-risk pregnant women.

The study was conducted using a randomized controlled trial design between April 1, 2024, and December 31, 2024, at a maternity hospital in Istanbul. A total of 100 high-risk pregnant women were randomized into two groups: 50 participants were assigned to the group receiving the holistic care program along with routine midwifery care (intervention), and 50 were assigned to the group receiving only routine midwifery care (control).

The Holistic Care Program for High-Risk Pregnancies consists of three sessions: Physiological Information and Preparation for High-Risk Pregnancy, Psychological Support and Preparation, and Creative Practices and Final Evaluation.

Research data were collected using five forms: Informed Consent Form, Demographic Information Form, Perceived Stress Scale for High-Risk Pregnancies Based on Neuman Systems Model, Brief Symptom Inventory, and Holistic Care Program Evaluation Form for High-Risk Pregnancies.

DETAILED DESCRIPTION:
Introduction: The presence of increased health risks or complications for either the mother, the fetus, or both during pregnancy or childbirth is referred to as high-risk pregnancy. Visual and socially enriched individualized educational programs for high-risk pregnancies are emerging as an essential component of providing holistic care that addresses medical and emotional needs. These educational programs aim to reduce stress and uncertainty that pregnant women may encounter during the perinatal period by helping them better understand their health conditions and the baby's condition. It is believed that individualized education provided to high-risk pregnant women receiving care in perinatology clinics can strengthen their stress-coping mechanisms and allow them to respond more effectively to emotional needs during this period.

Objective: This study aims to evaluate the effects of a holistic care program on the stress levels and mental health of high-risk pregnant women. In this context, the study seeks to explore the program's potential to enhance stress-coping mechanisms, positively influence mental health, and increase overall health awareness among high-risk pregnant women.

Methods: The study was conducted as a randomized controlled trial in the pregnancy follow-up outpatient clinic of a maternity hospital in Istanbul between April 1, 2024, and December 31, 2024. A total of 100 pregnant women were included in the study and randomly assigned to one of two groups:

Intervention Group: 50 participants Control Group: 50 participants Data were collected at two time points: a pre-test on the first day of group assignment and a post-test on the day of discharge. Research data were gathered through face-to-face interviews using five forms: Informed Consent Form, Demographic Information Form, Perceived Stress Scale for High-Risk Pregnancies Based on Neuman Systems Model, Brief Symptom Inventory, and Holistic Care Program Evaluation Form for High-Risk Pregnancies.

The intervention group received midwifery counseling and care accompanied by the Holistic Care Program for High-Risk Pregnancies. The control group received only the standard midwifery care provided by the clinic.

Intervention Group Applications: High-risk pregnant women admitted to the perinatology clinic and assigned to the intervention group participated in a Holistic Care Program for High-Risk Pregnancies in addition to the midwifery care provided at the clinic. The implementation of the program involved two phases: preparation and application.

Preparation Phase: The content of the Holistic Care Program for High-Risk Pregnancies, shaped by Neuman's Systems Model, was developed. Existing childbirth preparation programs and topics essential to high-risk pregnancy counseling were considered. Experts, including childbirth preparation instructors and academic midwifery professionals (2 Professors, 3 Associate Professors, 3 Assistant Professors, 2 Research Assistants, and 1 Lecturer), reviewed the program, and modifications were made based on their recommendations.

Application Phase: After finalizing the program content, the education sessions were scheduled. Sessions were held in a dedicated clinical space, taking into account clinical conditions, working schedules, and the treatment hours of the participants. The total program duration was planned for 6 hours and 15 minutes, delivered across three sessions and six meetings.

Session 1: Group education focused on physiological information and preparation from high-risk pregnancy to childbirth. This 2-hour session, conducted in two meetings, covered physiological aspects, body structures, and functions.

Session 2: Individual education focused on psychological support and preparation, aiming to enhance emotional resilience during pregnancy. This 2-hour session, conducted in two meetings, addressed psychological, sociocultural, and spiritual aspects of life.

Session 3: Group education titled "The Compassion of Hands: Bonding and Relaxation Techniques During Pregnancy" was conducted as a 2-hour and 15-minute session. This session focused on spiritual and emotional aspects, emphasizing bonding between the pregnant woman and her baby.

Control Group Applications: Routine midwifery care procedures followed in the perinatology clinic were applied to the control group.

Data Analysis: Data were analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0. Descriptive statistical analyses (frequency, percentage, minimum-maximum values, median, mean, and standard deviation) were employed. The suitability of data for normal distribution was tested using Kolmogorov-Smirnov and Shapiro-Wilk tests.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the study and over the age of 18,
* Ability to understand and speak Turkish,
* Being a primiparous woman,
* Being in the third trimester of pregnancy.
* Being hospitalized in the perinatology ward and receiving care for at least 3 days
* Having at least one diagnosed high-risk pregnancy condition

Exclusion Criteria:

* Not willing to participate in the study
* Presence of a fetal anomaly
* Risk of fetal loss
* Having previously received childbirth preparation education

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
"Perceived Stress Scale in High-Risk Pregnancies Based on the Neuman Systems Model (PSS-HRP-NSM)" | At the end of the 3-day holistic care program
  The scale consists of 34 items covering five life domains outlined in the Neuman Systems Model: physiological, psychological, sociocultural, developmental, and spiritual. It is a five-point Likert scale ranging from "Never (1)" to "Always (5)," with total scores ranging between 34 and 170. The sum of subscale scores reflects stress levels in the respective life domains, while the total score indicates overall stress levels. Items 22, 30, 31, 32, and 33 are reverse-coded. In the original study, the overall Cronbach's Alpha value was found to be 0.87, whereas, in this study, it was determined to be 0.954. Subscale Cronbach's Alpha values were calculated as 0.892 for the physiological domain, 0.911 for the psychological domain, and 0.867 for the sociocultural/developmental/spiritual domain. The scale was administered to both intervention and control groups as pre-test and post-test in this study, with higher scores indicating higher perceived stress levels in the respective life domains

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI) | At the end of the 3-day holistic care program
  The Brief Symptom Inventory (BSI), developed by Derogatis (1992), is a 53-item shortened version of the SCL-90-R, measuring psychological symptoms across five subscales: anxiety, depression, negative self-concept, somatization, and hostility. Responses are recorded on a 5-point Likert scale (0: Not at all, 4: Extremely), with higher scores indicating greater psychological distress. In the Turkish validation by Şahin et al. (2002), Cronbach's Alpha values ranged from 0.70 to 0.88, with an overall reliability of 0.94.
  In this study, the BSI showed an overall Cronbach's Alpha of 0.969. Subscale reliabilities were 0.869 for anxiety, 0.922 for depression, 0.900 for negative self-concept, 0.831 for somatization, and 0.844 for hostility. The scale was applied as both pre-test and post-test, with higher scores indicating increased psychological symptoms.

OTHER OUTCOMES:
Evaluation Form for the Holistic Care Program in High-Risk Pregnancies | At the end of the 3-day holistic care program
  This form, prepared by the researchers, begins with information about the participant's high-risk pregnancy process and hospitalization period, aiming to evaluate various aspects of the program. Elements such as the program's content, the appropriateness of the training duration, the effectiveness of the training services provided, and its contribution to stress management are thoroughly examined. Additionally, the educator's communication skills, adequacy in providing information and support, overall satisfaction level, and the program's impact on the hospitalization process are assessed. Participants were also asked to share the parts of the program they liked the most, the strengths of the counseling services, and suggestions for areas that need improvement. This form was completed by participants exclusively in the intervention group at the end of the training.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Uskudar Univercity, Istanbul, ümraniye
  - Üsküdar Üniversitesi, Istanbul, ümraniye

IPD SHARING:
Plan to Share IPD: Yes
The data requested by the researcher will be shared by the researcher in accordance with the confirmation of its intended use.
Supporting Information: CSR

REFERENCES:
- [Background] Carolan-Olah M, Sayakhot P. A randomized controlled trial of a web-based education intervention for women with gestational diabetes mellitus. Midwifery. 2019 Jan;68:39-47. doi: 10.1016/j.midw.2018.08.019. Epub 2018 Sep 5. PMID 30343264
- [Background] Schiele C, Goetz M, Hassdenteufel K, Muller M, Graf J, Zipfel S, Wallwiener S. Acceptance, experiences, and needs of hospitalized pregnant women toward an electronic mindfulness-based intervention: A pilot mixed-methods study. Front Psychiatry. 2022 Aug 22;13:939577. doi: 10.3389/fpsyt.2022.939577. eCollection 2022. PMID 36072461
- [Background] Anolak H, Lau F, Davis D, Browne J, Watt B. Creative arts intervention in support of women experiencing a high-risk pregnancy: A qualitative descriptive thematic analysis. Sex Reprod Healthc. 2023 Jun;36:100830. doi: 10.1016/j.srhc.2023.100830. Epub 2023 Mar 3. PMID 36898309